CLINICAL TRIAL: NCT05231551
Title: Using Embryo Organoids (i.e. Embryoids) to Discover Human-specific Mechanisms of Preimplantation Embryo Development and Early Pregnancy
Brief Title: Using Embryo Organoids to Discover Human-specific Mechanisms of Preimplantation Embryo Development and Early Pregnancy
Acronym: EMBRYOx
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0069
Record Dates: First submitted 2022-02-07; First posted 2022-02-09 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Infertility
Keywords: Embryo development; Implantation; Oxygen; Trophoblast organoid; In vitro fertilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissues of first-trimester human placentas after abortion donated to research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-group study: Patients having first trimester voluntary termination of pregnancy in Montpellier university hospital.
  Interventions: Procedure: Placental tissues

INTERVENTIONS:
Procedure: Placental tissues — Placental tissues are collected after aspiration of abortion products. They are treated immediately in order to isolate placental stem cells. Organoid culture is established and the obtained embryoids are cultured in monophasic or biphasic oxygen conditions. Extra organoids are cryopreserved in liquid nitrogen

SUMMARY:
EMBRYOx study aims to establish and validate the use of trophoblast organoids (embryoids) from trophoblast placental stem cells as a 3D research model in understanding further preimplantation embryo development in vitro. The organoids are capable of proliferation, differentiation, and implantation in a matrix, reproducing early human embryo development.

DETAILED DESCRIPTION:
Study objectives:

Our primary objective is to compare the transcriptomic profiles of embryoids with those obtained from human embryos donated to research and cultured in two different oxygen conditions (monophasic oxygen strategy: 5% of O2 for 5 days vs. biphasic oxygen strategy: 5% of O2 for 3 days and 2% of O2 afterwards for 2 days). The transcriptomic profiles of human embryos donated to research and cultured in two different oxygen conditions were obtained in our previous study (PMID: 34789773). The biphasic oxygen strategy turned out to be beneficial for early embryo development and pregnancy. The comparison of transcriptomic profiles could allow us to validate the embryoids as a model in the study of preimplantation embryo development in vitro. Moreover, this could permit us to better understand the molecular mechanisms associated with the positive impact of the biphasic oxygen conditions on embryo development.

Our secondary objective is to identify new non-invasive biomarkers predictive for preimplantation embryo development and pregnancy.

This is a prospective, monocentric, observational study.

Study population:

Patients having first trimester voluntary termination of pregnancy in Montpellier University Hospital which have previously signed an informed consent. Placental tissues are collected after aspiration of abortion products. At least 5 organoids populations from 5 different placentas will be generated.

Material and methods:

* Collection of placental tissues after first trimester voluntary termination of pregnancy. Foetal tissues will not be collected as organoids are formed exclusively of trophoblast placental stem cells.
* Isolation of trophoblast placental stem cells.
* Culture, differentiation, and formation of embryoids.
* Culture of embryoids under monophasic (5% of O2 for 5 days) or biphasic oxygen conditions (5% of O2 for 3 days and 2% of O2 after for 2 days).
* ARN extraction (MiniKit Qiagen) and establishment of transcriptomic profiles (MGX-Montpellier GenomiX platform).
* Comparison of the transcriptomic profiles obtained with those of human embryos (Ingenuity Pathway Analysis).
* Cryopreservation of extra organoids in liquid nitrogen.

Assessment criteria:

Embryoids' dimension (100-150 um), proliferation/apoptosis index, expression of trophoblast markers (GATA3, KRT7, EGFR, TFAP2A, TFAP2C) by qPCR (Affymetrix Clariom) or immunohistochemistry.

Results and perspectives:

The investigators are expecting to obtain higher expression of proliferation, cellular survivor and pluripotency genes in embryoids cultured in biphasic oxygen conditions. If the investigators find the same outcomes after transcriptomic analysis of trophoblast organoids as those of human embryos, this would support the utilisation of organoids as a model in the study of human preimplantation embryo development.

Subsequently, the investigators could test the impact of other factors on the organoids' development (as culture medium composition, pH, etc.) and optimise the predictive value of non-invasive biomarkers (cf-DNA, PROK1 etc.).

ELIGIBILITY:
Inclusion criteria:

- No smoking patients without drug consumption or previous medication who are having first trimester voluntary termination of pregnancy surgically or medically induced.

Exclusion criteria:

- Patients smoking, drug consumption, previous medication

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients having first trimester voluntary termination of pregnancy in Montpellier university hospital which have previously signed an informed consent. Placental tissues are collected after aspiration of abortion products.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of research in preimplantation embryo development in vitro | 1 day
  Establish and validate the use of embryoids from trophoblast placental stem cells as a 3D model for research in preimplantation embryo development in vitro.Our primary objective is to compare the transcriptomic profiles of embryoids with those obtained from human embryos donated to research and cultured in two different oxygen conditions (monophasic oxygen strategy: 5% of O2 for 5 days vs. biphasic oxygen strategy: 5% of O2 for 3 days and 2% of O2 afterwards for 2 days). The transcriptomic profiles of human embryos donated to research and cultured in two different oxygen conditions were obtained in our previous study (PMID: 34789773). The biphasic oxygen strategy turned out to be beneficial for early embryo development and pregnancy.

SECONDARY OUTCOMES:
Rate of Identification of new non-invasive biomarkers | 1 day
  Identification of new non-invasive biomarkers which are predictive for preimplantation embryo development and pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Samir HAMAMAH, PUPH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC